CLINICAL TRIAL: NCT05317429
Title: Measuring Postprandial Glycaemic Responses to Carbohydrate-rich Meals Using a Standardised Remote Monitoring Protocol
Brief Title: Glycaemic Responses to Carbohydrate-rich Meals (GlyCarb)
Acronym: GlyCarb
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Quadram Institute Bioscience (Other)
Collaborators: Norfolk and Norwich University Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: QIB07/2020
Record Dates: First submitted 2022-02-16; First posted 2022-04-07 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Glycaemia
Keywords: Carbohydrates; Starch
MeSH Terms: interventions — Carbohydrates

STUDY DESIGN:
Intervention Model Description: Randomised crossover study
Who Masked: Investigator, Outcomes Assessor
Masking Description: Blinding will be conducted by a member of staff who is independent of the study team. For all studies, an effort will be made to blind the research team and study participants to the test and reference meals. Whilst we recognize that this approach is 'gold standard' it may not be possible in all circumstances, for example due to the different appearance of some food products.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): Carbohydrate-rich meal
  Interventions: Other: A meal delivering 75 g of carbohydrate
- Control (Active Comparator): Carbohydrate-rich meal
  Interventions: Other: A meal delivering 75 g of carbohydrate

INTERVENTIONS:
Other: A meal delivering 75 g of carbohydrate — The nature of the test meal will depend upon the research question being addressed and it is anticipated that the test meals may include (but are not limited to) the following:
  (i) Re-structured, enriched, and/or reformulated or non-conventionally processed food products (ii) Model food matrices with different structures or types of carbohydrate e.g. soups with different viscosity.

SUMMARY:
Carbohydrate-rich foods such as potatoes, bread, rice, pasta, breakfast cereals, biscuits and other snacks are a major component of the human diet. The effect of different carbohydrate-rich foods on blood sugar (glucose) levels after a meal varies between foods. This is relevant to health because studies have shown that regular intake of carbohydrate foods that cause large increases in blood glucose levels after ingestion can be detrimental to metabolic health.

The aim of the GlyCarb study is to investigate how food structure influences postprandial glycaemic responses to carbohydrate foods.

This will be achieved through a series of acute postprandial studies (up to 5 studies), wherein healthy participants within each postprandial study consume a pair of carbohydrate-rich test meals while wearing a continuous glucose monitoring system (CGM).

Each postprandial study will use the same GlyCarb Remote standard protocol, where a randomised cross-over design is used to measure the glycaemic response to two carbohydrate-rich test meals, one "test" and one "control". Both meals will be matched by carbohydrate content, contain similar ingredients and have a similar physical appearance, but will differ in one key food property (e.g., altered food structure) to test its effect on postprandial glycaemia.

In each postprandial study, habitual dietary intake and body composition will be captured at baseline as part of the participant characterisation. Participants will consume two different carbohydrate-rich test meals twice, on separate occasions, in a randomly allocated order over a 10 to 14-day period of continuous glucose monitoring. Data from the continuous glucose monitors will be used to assess the postprandial glycaemic response to each carbohydrate food. The participants will be required to complete brief questionnaires designed to evaluate differences in palatability (taste, texture, portion size) and satiety amongst test meals. Study participant feedback will be requested at the end of the study and used to assess and improve future study procedures.

The GlyCarb study will enable new understanding of how food properties influence glycaemic responses to different types of carbohydrate foods. Ultimately, the findings will inform the rational design or reformulation of food products and diets to support a healthy glucose metabolism.

DETAILED DESCRIPTION:
The overarching aim of this project is to investigate a wide range of carbohydrate rich test meals (from 'off the shelf' commercially available products, through to enriched, restructured and re-formulated food products) on postprandial glycaemic response in normo-glycaemic individuals.

The 'remote' study protocol has been designed to maintain social distancing and thereby reduce risk of COVID19 transmission between participants and researchers during the ongoing outbreak. It also makes excellent use of continuous glucose monitoring devices, which enable continuous recording of participant body sugar levels in 'free-living' conditions. At no point will the participant be required to attend a clinical research facility. Support from the study team to participants will be provided through virtual appointments.

The study population will be healthy participants. Participants will also need to have access to a smart phone to be used in conjunction with the CGM as well as for virtual study appointments (video call) and to complete online forms.

The precise test meals will vary from study to study, and will always need to meet a set standard with regard to microbiological safety, traceability and nutrient composition. As an extra precaution, participants with ANY food allergy will not be able to take part in the study. The meals will be well characterised and details of nutrient composition, ingredients, allergens etc. will be provided to participants prior to consent.

Informed consent - to ensure participants can make an informed decision as to whether or not they wish to take part on the trial they will be provided with a study specific PIS and invited to participate in an informal discussion about the study. Consent will be obtained by a member of staff who is GCP trained and experienced in conducting human intervention trials. In line with the 'remote' nature of the study, participants and study team members will be video and audio recorded during the consent procedure, with their permission. Hard copies of the consent form will also be initialled and signed by the participant and countersigned by the study team as written informed consent.

Risks/Burdens - (i) At the eligibility assessment a small blood sample is collected. Participants may feel a little discomfort on initial insertion of the needle or bruising at the site of venepuncture. Similarly, there may be some discomfort during finger prick testing. (ii) The CGM sensor may be secured by an adhesive 'plaster' which could cause irritation. Should this occur the CGM could be secured in place with an elastic support bandage such as tubigrip or similar.

iii) This study involves periods of fasting. Participants will be advised to drink water during the fasting period. All study sessions will be scheduled for the morning time to reduce the length of fast.

(iv) As part of the eligibility assessment it is possible that some test results are returned as abnormal. Abnormal blood and urine test results are reviewed by our medical doctor who advises whether inclusion, re-screen or exclusion is appropriate. In addition, copies of all test results (whether abnormal or not) will be sent to the participants GP.

Participants will complete a Food Frequency Questionnaire to capture the habitual diet as a baseline characteristic as well as measure fat and muscle mass using a smart scale.

Data protection and confidentiality - Participants will be assigned a unique code and a Quadram Institute Bioscience (QIB)-based email which will be used on all samples/data arising from a study. Paper documents containing identifiable information (e.g. consent forms) and coded information will be kept in locked cabinets at the QIB. The file linking the code with the participant will be kept separately. All documents will only be accessible to the members of the study team. All electronic data will be stored on a password protected shared file at the QIB and access will be limited to members of the study team.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥ 18 years of age
* Have access to/own a smartphone or tablet or computer and are willing to use this with apps needed for the study
* BMI between 18 and 30 kg/m2 (calculated from self-reported height and weight)
* Fasted HbA1C < 42 mmol/mol (6.0%)
* Willing to consume study foods (study foods and ingredients are discussed during the study talk)

Exclusion Criteria:

* Smokers of tobacco-based cigarettes or electronic cigarettes (or stopped smoking less than 6 months ago)
* Gastro-intestinal disease/disorders e.g., Crohn's disease/ulcerative colitis
* Other medical conditions that are judged to affect the study outcome or which may compromise the well-being of the participant e.g., active cancer, haemophilia. This will be assessed on a case-by-case basis.
* Type 1 diabetes or insulin-dependent or non-insulin-dependent type 2 diabetes
* Active infection with COVID-19, unless they are willing to postpone the screening until after the end of the self-isolation period (10 days from test or symptoms).
* Prescribed and non-prescribed medications that may affect the study outcome or which may compromise the well-being of the participant e.g., warfarin, proton-pump inhibitors. This will be assessed on a case by-case-basis.
* Dietary supplements that are judged to affect the study outcome unless the participant is willing to discontinue them for 4 weeks preceding the start of the study and for the duration of the study. This will be assessed on a case-by-case basis and includes protein supplements (shakes) or supplements that are not taken on a regular basis (on and off), particularly those containing ascorbic acid which may affect glucose readings.
* Any known allergy, intolerance, or sensitivity to any food products oradhesives (for CGM application).
* Those following a restrictive diet that may affect the study outcome (e.g., 5:2 diet) unless they are willing to suspend the diet for the duration of the study.
* Women who are, or have been pregnant, within the last 12 months or who are breast-feeding
* Parallel participation in another research project that involves dietary intervention.
* Any person related to or living with any member of the study team.
* Those who are part of the line manager/supervisory team of the Chief Investigator
* Lack of capacity to provide written informed consent.
* Clinical eligibility test results deemed by the CRF medical advisor to be indicative of a health problem which may compromise the well-being of the participant or which could affect the study outcome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2022-02-14 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Fasting and postprandial glucose levels measured in interstitial fluid | 0-4 hours after the test meal
  Maximum rise in glucose concentration from fasted levels (iCmax)

SECONDARY OUTCOMES:
Glycaemic response indicators | 2 to 4 hours after the test meal
  Incremental area under the curve (iAUC) for the first peak
Glycaemic response indicators | 2 to 4 hours after the test meal
  Incremental area under the curve (iAUC) between 0-120 min
Glycaemic response indicators | 2 to 4 hours after the test meal
  Minimum glucose concentration (Cmin)
Glycaemic response indicators | 2 to 4 hours after the test meal
  Time to reach glucose peak concentration (Tmax), time to reach minimum concentration (Tmin)
Glycaemic response indicators | 2 to 4 hours after the test meal
  Time to reach minimum glucose concentration (Tmin)
Glycaemic response indicators | Over 14 days
  Coefficient of variation (CV)
Glycaemic response indicators | Over 14 days
  Time in Range (TIR)
Glycaemic response indicators | Over 14 days
  Mean Amplitude Glucose Excursion (MAGE)
Glycaemic response indicators | Over 14 days
  Mean of daily differences (MODD)
Satiety | Time 0 (before meal), 30 (after meal), 60, 120, 180 and 240 minutes after each test meal.
  Online survey responses from participants.
Palatability | Once per day on intervention days, four times per study
  Online survey responses from participants. Palatability scores (recorded once after each test meal), from 'Dislike Very Much' to 'Like Very Much'.

OTHER OUTCOMES:
BMI | Baseline
  weight and height will be combined to report BMI in kg/m^2
Body composition | Baseline
  Percentage of fat mass
Body composition | Baseline
  Percentage of muscle mass
Habitual dietary Intake | Baseline
  Food Frequency Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Cathrina Edwards, PhD, Principal Investigator — Quadram Institute Bioscience
Locations (1):
- Quadram Institute, Norwich, Norfolk, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for primary and secondary outcome measures will be made available
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available after publication in scientific journal within 18 months of study completion
Access Criteria: Data access will be reviewed by the study team